CLINICAL TRIAL: NCT01810549
Title: Role of Interleukin-1 in Postprandial Fatigue - The Cheesecake Study. A Randomized, Double-blind, Single Dose of Anakinra, Placebo-controlled, Cross-over Proof-of-concept Study.
Brief Title: Role of Interleukin-1 in Postprandial Fatigue - The Cheesecake Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: EK 303/12
Record Dates: First submitted 2013-03-04; First posted 2013-03-13 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2013-03

CONDITIONS: Postprandial Fatigue
Keywords: Fatigue
MeSH Terms: conditions — Fatigue | interventions — Interleukin 1 Receptor Antagonist Protein; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anakinra (Active Comparator): Anakinra 100mg. Every subject will receive one subcutaneous injection of study drug once during the study, a total of one injection.
  Interventions: Drug: Anakinra
- Placebo (Placebo Comparator): Every study participant will receive a single subcutaneous injection of Placebo once during the study, a total of one injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anakinra — Each subject will receive one single subcutaneous injection of 100mg Anakinra during the study, a total of one injection.
  Other Names: Kineret
  Arms: Anakinra
Drug: Placebo — Every subject will receive one single subcutaneous injection of Placebo during the study, a total of one injection.
  Other Names: Saline
  Arms: Placebo

SUMMARY:
The aim of the study is to investigate, if postprandial fatigue symptoms after ingestion of a high-fat, high-carbohydrate meal are regulated by Interleukin (IL)-1 and can be prevented by inhibition of IL-1 using a single dose injection of a specific IL-1 receptor antagonist.

ELIGIBILITY:
Inclusion Criteria:

* male
* non-smoking
* apparently healthy
* BMI >18 and ≤25 kg/m2
* Age 20-50 years
* Willingness to use contraceptive measures adequate to prevent the subject's partner from becoming pregnant during the study. Adequate contraceptive measures include hormonal methods used for two or more cycles prior to screening (e.g., oral contraceptive pills, contraceptive patch, or contraceptive vaginal ring), double barrier methods (e.g., contraceptive sponge, diaphragm used in conjunction with contraceptive foam or jelly, and condom used in conjunction with contraceptive foam or jelly), intrauterine methods (IUD), sterilization (e.g., tubal ligation or a monogamous relationship with a vasectomized partner), and abstinence.

Exclusion Criteria:

* Clinical signs of infection in the week before inclusion or history of infection during the last 2 months (CRP >5mg/l)
* Impaired fasting glucose (fasting plasma glucose >5.5mmol/l)
* Hematologic disease (leukocyte count < 1.5x109/l, hemoglobin <11 g/dl, platelets <100 x 103/ul)
* Kidney disease (creatinine > 1.5 mg/dL))
* Liver disease (transaminases >2x upper normal range)
* Heart disease
* Pulmonary disease
* Inflammatory disease
* History of carcinoma
* History of tuberculosis
* Alcohol consumption >40g/d
* Smoking
* Known allergy towards Anakinra
* Known allergy towards ingredients of the test meal
* Current treatment with any drug in the week before inclusion, including vitamin supplementation (especially vitamin C and E)
* Use of any investigational drug within 30 days prior to enrollment or within 5 half-lives of the investigational drug, whichever is longer
* Subject refusing or unable to give written informed consent

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Postprandial fatigue | pre-study drug (180 minutes pre-meal), 30 minutes pre-meal and 30 minutes post-meal
  Fatigue will be assessed using the Fatigue Scale for Motor and Cognitive Functions (FSMC) pre-study drug (means 180 minutes before ingestion of the test meal), 30 minutes before ingestion of the test meal and again 30 minutes after ingestion of the test meal. The outcome measure for which data will be presented is the change in fatigue measured 30 minutes before and 30 minutes after ingestion of the test meal in participants receiving kineret vs. placebo. Fatigue will also be assessed before administration of the study drug (180 minutes before test meal) to unravel a possible influence of the study drug itself on fatigue symptoms.

SECONDARY OUTCOMES:
Postprandial depression | pre-study drug (180 minutes pre test meal), 30 minutes pre-meal, 30 minutes post-meal
  Depression will be assessed using the Hospitality Anxiety and Depression Scale - german version (HADS-D) pre-study drug (means 180 minutes before ingestion of the test meal), 30 minutes before ingestion of the test meal and again 30 minutes after ingestion of the test meal. The outcome measure for which data will be presented is the change in depression measured 30 minutes before and 30 minutes after ingestion of the test meal in participants receiving kineret vs. placebo. Depression will also be assessed before administration of the study drug (180 minutes before test meal) to unravel a possible influence of the study drug itself on depression.
Postprandial cognitive processing speed | pre-study drug (180 minutes before test meal), 30 minutes pre-meal, 30 minutes post-meal
  Cognitive processing speed will be assessed using the oral version of the Symbol Digit Modalities Test (SDMT) version A before study drug (means 180 minutes before ingestion of the test meal), version B 30 minutes before ingestion of the test meal and version A 30 minutes after ingestion of the test meal. The outcome measure for which data will be presented is the change in cognitive processing speed measured 30 minutes before and 30 minutes after ingestion of the test meal in participants receiving kineret vs. placebo. Cognitive processing speed will also be assessed before administration of the study drug (180 minutes before test meal) to unravel a possible influence of the study drug itself on depression. Version A and B will be used alternately to prevent a learning effect in this test.
Insulin, C-peptide, Glucose | -180, -10 and 0 minutes before ingestion of the test meal; 5, 15, 30, 60, 90, 120, 180 and 240 minutes after full ingestion of the test meal
Gut hormones and inflammatory markers | -180, -10 and 0 minutes before ingestion of the test meal; 5, 15, 30, 60, 90, 120, 180 and 240 minutes after full ingestion of the test meal

CONTACTS AND LOCATIONS:
Overall Officials: Marc Y Donath, Prof., Principal Investigator — Univesity Hospital Basel
Locations (1):
- University Hospital Basel, Basel, Switzerland